CLINICAL TRIAL: NCT03699878
Title: Impact of Perioperative Shedding of the Endothelial Glycocalyx on Short-term Postoperative Complication in Patients Undergoing Robot-assisted Esophagectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0773
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Robotic Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing robotic esophagectomy: Patients 20 years or older who undergo robotic esophagectomy

SUMMARY:
The aim of this study was to determine whether changes in serum levels of syndecan-1 before and after surgery, which is an index related to injury of the endothelial glycocalyx layer, are associated with postoperative short-term complications and mortality in patients undergoing robotic esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

1. patients 20 years or older who undergo robotic esophagectomy

Exclusion Criteria:

1. Emergency surgery
2. If the subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)
3. Chronic kidney disease (eGFR <30 mL / min / 1.73 m2)
4. Pregnant and lactating women
5. Use of oral anticoagulants

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients 20 years or older who undergo robotic esophagectomy
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
base blood concentration of syndecan-1 | within 1 hour before surgery
  preoperative baseline serum levels of syndecan-1
blood concentration of syndecan-1 at the end of the surgery | within 5 minutes after the end of surgery (when thd surgical drape is removed)
  blood concentration of syndecan-1 at the end of the surgery
blood concentration of syndecan-1 at 24 hours after surgery | 24 hours after the end of surgery
  blood concentration of syndecan-1 at 24 hours after surgery

SECONDARY OUTCOMES:
Unanticipated Post-Operative Invasive Procedure (STS GTSD 2.41 #3330) | during this 1 day hospital visit.
  Indicate if the patient had an unplanned invasive procedure after surgery. Examples includes return to the operating room for a redo surgical procedure, a percutaneous procedure performed at bedside or in the radiology suite, a tracheostomy, and wound opening at bedside. Exclusions: postoperative toilet bronchoscopy, central venous access, arterial line placement, foley catheter placement.
Anastomotic leak following esophageal surgery(STS GTSD 2.41 #3350) | within 30days after end of surgery
  Indicate if the patient had an anastomotic leak following esophageal surgery.
Respiratory Failure(STS GTSD 2.41 #3480) | within 30days after end of surgery
  Indicate whether the patient experienced respiratory failure in the postoperative period requiring mechanical ventilation and/or reintubation.
initial ventilatory support greater than 48 hours (STS GTSD 2.41 #3520) | within 30days after end of surgery
  Indicate if the patient initially was ventilated greater than 48 hours in the postoperative period. If the patient is reintubated, select the postoperative event "Respiratory Failure" and do not select this element even if the reintubation ventilator support is > 48 hours. Ventilator support ends with the removal of the endotracheal tube or if the patient has a tracheostomy tube, until no longer ventilator dependent.
pneumonia (STS GTSD 2.41 #3460) | within 30days after end of surgery
  Indicate if the patient experienced pneumonia in the postoperative period. Pneumonia is defined as meeting three of five characteristics: fever (> 100.4 F or 38 C), leukocytosis, CXR with infiltrate, positive culture from sputum, or treatment with antibiotics.
renal failure(STS GTSD 2.41 #3810) | within 30days after end of surgery
  Indicate whether the patient had acute renal failure or worsening renal function resulting in any of the following:
  1. New requirement for dialysis post-operatively
  2. Increase in serum creatinine level 3.0 x greater than baseline
  3. serum creatinine level ≥4 mg/dL , with an acute rise of at least 0.5 mg/dl
mortality(Status 30 Days after Surgery, STS GTSD 2.41 #3950) | 30days post-surgery
  Indicate whether the patient was alive or dead at 30 days post-surgery (whether in the hospital or not).
  time frame: 30days post-surgery
Acute kidney injury | within 48 h after end of surgery
  defined as an absolute increase in serum creatinine level C0.3 mg/dL, a 50% (1.5-fold) increase in serum creatinine level from baseline, or a reduction in urine output (documented oliguria< 0.5 mL/kg/h for 6h)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided